CLINICAL TRIAL: NCT02014363
Title: Double Blind, Non-inferiority Study to Evaluate the Antidepressant Activity of ETS6103 Compared to Amitriptyline in Treating Major Depressive Disorder in Patients With Unsatisfactory Response to Selective Serotonin Re-uptake Inhibitors.
Brief Title: Safety and Efficacy Study Comparing ETS6103 With Amitriptyline in the Treatment of Major Depressive Disorder (MDD)
Acronym: ETS6103-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: e-Therapeutics PLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ETS6103-003; 2013-000719-26 (EudraCT Number)
Record Dates: First submitted 2013-12-12; First posted 2013-12-18 (Estimated); Results first posted 2017-01-11 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2016-11

CONDITIONS: Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Amitriptyline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- ETS6103 (low dose) (Experimental): ETS6103 (low dose) extended release tablets (encapsulated) taken once daily orally for the duration of randomised phase of the study (8 weeks).
  Interventions: Drug: ETS6103 (low dose)
- ETS6103 (high dose) (Experimental): ETS6103 (high dose) extended release tablets (encapsulated) taken once daily orally for the duration of randomised phase of the study (8 weeks).
  Interventions: Drug: ETS6103 (high dose)
- Amitriptyline (Active Comparator): Amitriptyline tablets (encapsulated) Standard dosing regime
  Interventions: Drug: Amitriptyline
- Lead-in phase (No Intervention): Citalopram tablets:
  Standard dosing regime

INTERVENTIONS:
Drug: ETS6103 (low dose)
  Arms: ETS6103 (low dose)
Drug: ETS6103 (high dose)
  Arms: ETS6103 (high dose)
Drug: Amitriptyline
  Arms: Amitriptyline

SUMMARY:
To demonstrate that the antidepressant activity of ETS6103 is not inferior to amitriptyline in subjects who have an unsatisfactory response to / are resistant to treatment with SSRIs.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Male or female
* Age 18-65 years inclusive
* Subjects with a current episode of moderate to severe Major Depressive Disorder meeting the criteria of Diagnostic and Statistical Manual of Mental Disorders (DSM) IV -TR and documented using the brief structured interview Mini International Neuropsychiatric Interview (MINI) version 5.0 and with a minimum duration of two weeks and a maximum of twelve months
* Minimum Hamilton Depression Scale (HAM-D) 17 items total score of 18 at screening and ≥12 at the end of the lead-in phase prior to randomization.
* Female subjects of childbearing potential must have a negative pregnancy test at the Screening Visit and must use an acceptable method of contraception throughout the study and for 30 days after. Male subjects with female partners of child-bearing potential must use an acceptable method of contraception throughout the study and for 30 days after.
* Able to understand and comply with the requirements of the study as judged by the investigator

Exclusion Criteria:

* Considered by the investigator to be at significant risk of suicide or scoring 5 or more on the Montgomery Asberg Depression Rating Scale (c) question 10
* Significant other psychiatric illness which would interfere with trial assessments co-morbid generalized anxiety disorder (GAD) and panic disorder will be permitted where MDD is considered the primary diagnosis
* Significant physical illness which would interfere with trial assessments
* Recent (within 1 week of screening) antidepressants (except for fluoxetine [within 4 weeks of screening] and St John's Wort or Monoamine oxidase inhibitors (MAOI) [within 14 days of screening]),
* Benzodiazepine or any other psychotropic medication including lithium or other mood stabilizers within 1 week of screening
* Oral anticoagulant therapy within one month of screening
* Formal psychotherapy or alternative treatments for one week prior to screening or during the study
* Reduced hepatic function defined as liver enzyme levels ≥2.5 times upper limit of normal
* Renal insufficiency defined as creatinine clearance <30 mL/min
* Epilepsy
* Uncontrolled hypothyroidism
* Uncontrolled hypertension
* Acute porphyria
* Urinary retention, prostatic hypertrophy, narrow angle glaucoma or increased intraocular pressure or any other clinically relevant contraindication stated in the Summary of Product Characteristics (SmPC) for citalopram, tramadol or amitriptyline
* History of significant cardiac dysrhythmia or history of myocardial infarction within 1 year prior to screening
* Significant history of alcohol or substance abuse
* Regular alcohol intake above the recommended United Kingdom (UK) guideline of 4 units per day for males or 3 units per day for females
* Pregnant or lactating women
* Known hepatitis B or C or human immunodeficiency virus (HIV) or syphilis seropositivity.
* A corrected QT interval of >470ms for female subjects of >450ms for male subjects, calculated using the QTcB (Bazett Correction Formula) , or second degree or higher heart block on an electrocardiography (ECG) recording, at screening.
* Allergy to the study drugs or excipients
* Treatment with another investigational medicinal product within the 30 days prior to screening.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Actual)
Dates: Start 2013-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Alan G Wade, MBChb, Principal Investigator — CPS Research
Locations (1):
- CPS Research, Glasgow, Scotland, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- ETS6103 (Low Dose): ETS6103 (low dose) extended release tablets (encapsulated) taken once daily orally for the duration of randomised phase of the study (8 weeks).
  ETS6103 (low dose)
- ETS6103 (High Dose): ETS6103 (high dose) extended release tablets (encapsulated) taken once daily orally for the duration of randomised phase of the study (8 weeks).
  ETS6103 (high dose)
- Amitriptyline: Amitriptyline tablets (encapsulated) Standard dosing regime
  Amitriptyline
Period: Overall Study
Arm/Group | ETS6103 (Low Dose) | ETS6103 (High Dose) | Amitriptyline
Started | 55 | 54 | 55
Completed | 38 | 35 | 31
Not Completed | 17 | 19 | 24

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ETS6103 (Low Dose) | ETS6103 (High Dose) | Amitriptyline | Total
Number analyzed (Participants) | 55 | 54 | 55 | 164
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 55 | 54 | 55 | 164
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (11.85) | 41.1 (12.74) | 35.6 (11.95) | 38.8 (12.18)
Gender [Count of Participants; unit: Participants]
  Female | 16 | 14 | 19 | 49
  Male | 39 | 40 | 36 | 115
Region of Enrollment [Count of Participants; unit: Participants]
  United Kingdom | 55 | 54 | 55 | 164

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Baseline-adjusted (Montgomery-Asberg Depression Scale) MADRS Score at the End of Treatment.
Description: The mean difference in baseline-adjusted MADRS score at the end of treatment in the per protocol population using the last observation carried forward (LOCF) method. MADRS is used to assess the range of symptoms that are most frequently observed in patients with major depression. The MADRS test includes 10 items and uses a 0 to 6 severity scale, with higher scores indicating increasing depressive symptoms. The total MADRS score is derived by adding all the scores from the 10 items, meaning the lowest possible score is 0 and the highest possible is 60.
Time Frame: Baseline (start of randomized treatment) and 8 weeks post start of treatment
Population: Per protocol population (all subjects of the full analysis set for whom no relevant protocol deviations were documented).
Measure: Least Squares Mean (Standard Error); unit: Scores on a scale
Arm/Group | ETS6103 (Low Dose) | ETS6103 (High Dose) | Amitriptyline
Number analyzed (Participants) | 44 | 43 | 39
Scores on a scale | -6.1396 (1.64423) | -6.0076 (1.65174) | -11.3762 (1.7344)

ADVERSE EVENTS:
Arm/Group | ETS6103 (Low Dose) | ETS6103 (High Dose) | Amitriptyline
Serious Adverse Events (participants affected / at risk) | 1/55 | 1/54 | 1/55
Other Adverse Events (participants affected / at risk) | 43/55 | 50/54 | 47/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETS6103 (Low Dose) (N=55) | ETS6103 (High Dose) (N=54) | Amitriptyline (N=55)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ETS6103 (Low Dose) (N=55) | ETS6103 (High Dose) (N=54) | Amitriptyline (N=55)
Dry mouth (Gastrointestinal disorders) | 3 (3) | 7 (7) | 26 (26)
Vomiting (Gastrointestinal disorders) | 3 (4) | 6 (8) | 6 (6)
Nausea (Gastrointestinal disorders) | 6 (6) | 5 (7) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 3 (3) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 0 (0) | 2 (2) | 4 (4)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 5 (5)
Gastro-oesophageal reflux disease (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
Abnormal dreams (Psychiatric disorders) | 7 (7) | 8 (8) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 1 (1) | 5 (5)
Nightmare (Psychiatric disorders) | 2 (2) | 4 (4) | 1 (1)
Irritability (Psychiatric disorders) | 1 (1) | 2 (2) | 1 (1)
Headache (Nervous system disorders) | 6 (6) | 5 (5) | 3 (3)
Dizziness (Nervous system disorders) | 2 (2) | 5 (5) | 4 (4)
Tremor (Nervous system disorders) | 0 (0) | 0 (0) | 8 (8)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 5 (5)
Pruritus (Skin and subcutaneous tissue disorders) | 3 (3) | 7 (8) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 (4) | 1 (1) | 2 (2)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 5 (6) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 4 (4) | 5 (5) | 0 (0)
Fatigue (General disorders) | 3 (3) | 7 (7) | 4 (4)
Electrocardiogram QT prolonged (Investigations) | 3 (3) | 1 (1) | 2 (2)
Blood pressure increased (Investigations) | 0 (0) | 1 (1) | 3 (3)
Mean cell volume (Investigations) | 1 (1) | 2 (2) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 3 (3) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 2 (2) | 0 (0) | 3 (3)
Proteinuria (Renal and urinary disorders) | 1 (1) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
There is an agreement between the Principal Investigators and the Sponsor (or its agents) that restricts the PI's rights to discuss or publish trial results after the trial is completed.